CLINICAL TRIAL: NCT07391150
Title: Pilot Evaluation of 3D Designed Custom-made Integrated Mask/Headgear For Children Using Non-Invasive Ventilation (The "COMFORT" Study - Customised Masks For Overnight Respiratory Therapy)
Brief Title: NIV Mask and Headgear Evaluation
Acronym: NIV Masks
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other); University of Nottingham (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCH-2757
Record Dates: First submitted 2025-04-30; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIV Masks (Experimental)
  Interventions: Device: NIV Mask

INTERVENTIONS:
Device: NIV Mask — NIV Mask (custom)

SUMMARY:
Non-invasive ventilation (NIV) is the delivery of breathing support via a facemask. It is used to treat people whose natural breathing is ineffective. Evidence shows that, when used long-term, it improves both quality of life and life expectancy.

Ventilation is delivered in the home through a mask covering the nose or the nose and mouth. A good fit between the mask and the patient's face is essential to deliver the treatment effectively. Mass-produced masks are available for the adult market but in children it is often difficult to find a mask that provides an adequate fit. A particularly disadvantaged group is children with facial deformities or facial asymmetry. In these groups NIV may not be possible due to unavailability of an adequate mask.

Currently the options for these groups of children are to ventilate invasively via a breathing tube (tracheostomy) which can lead to serious complications and costly care-packages or to abandon ventilation, eventually leading to respiratory failure and premature death. Persevering with an inadequately fitting mask leads to pressure sores, impairment of facial bone growth and significant disturbance to the sleep of the child and family due to noise from air leakage from the mask and alarms from the ventilator. These problems lead to an increased burden on nursing and hospital resources as well as harm and suffering to patients.

The COMFORT study was funded by the NIHR in 2015 to develop novel mask-face interfaces to optimise mask fit to the needs of individual patients using 3D assessment and manufacturing technologies. Since then, we have developed a mask prototype and a modular headgear prototype that straps the mask onto the face. We have already demonstrated that our proposed method is more effective than a standard mass-produced mask/headgear in the laboratory setting with adult volunteers.

In the first part of this project, we will carry out a proof-of-concept study to test the prototype mask/headgear system with children and young people that currently use NIV but have a poorly-fitting mask. We will compare our new system with their current mask by asking them to rate them in terms of comfort and fit as well as measuring the effectiveness of their ventilation. In the second part, we will work with Imperial University, who have developed software to automate and speed up the manufacturing process. We will scan 120 children to help develop the software to be suitable for children and then repeat the proof-of-concept study with a mask manufactured using the automated process. Following these studies we will apply for funding to carry out a multicentre UK-wide clinical trial.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is a method of providing artificial respiratory support without placement of a tube in the airway; the air pressure is applied externally through the nose and/or the mouth. NIV was developed in the 1980s to support breathing in children with nocturnal hypoventilation due to neuromuscular weakness. In recent years the use of NIV has been offered to an extended group of patients with acute and chronic respiratory failure.

The aims of NIV are to improve gas exchange and to improve respiratory symptoms. Without ventilation, these patients will suffer chronic hypoxia resulting in pulmonary hypertension, cor pulmonale and premature death. NIV is effective in correcting nocturnal hypoventilation and in alleviating the associated symptoms. There is evidence that the use of NIV improves the quality of life in children with neuromuscular disorders and the life expectancy with those who decline NIV being more likely to die of respiratory failure within 2 years (6-12). NIV has been shown to reduce both hospital admissions (2-4 per year pre-NIV and 1 per year post-NIV) and days spent in hospital (40-50 per year pre-NIV and 10 per year post-NIV). Further work to look at this is underway within our group.

The biggest challenge with NIV treatment is enabling the child to tolerate the interface; the biggest cause of failure of NIV is the inability to fit a comfortable mask. Air leaks around the mask due to poor fit are a common reason for NIV to be ineffective and to be poorly tolerated. Pressure from an NIV mask on the growing face can result in under-development of the maxilla, leading to mid-face flattening and mal-occlusion of the teeth after as little as 4 weeks. Breakdown of the skin and pressure sores, usually on the bridge of the nose or forehead can occur when using mask ventilation. Prevention is better than cure and can be achieved if a suitably fitting mask is available.

NIV masks are available commercially for standard-size adults and children, but a good fit can be difficult to obtain in children with facial dysmorphic syndromes and other underlying co-morbidities. Custom-made masks are associated with a lower incidence of skin injury but are not available in most UK centres. The COMFORT project has developed a prototype custom made mask as well as a modular headgear prototype using 3D scanning and printing technology. Further work is taking place to inform the optimal 3D scanning technique and a software algorithm to automate the design process. This pilot clinical study will gain data in order to inform a multicentre clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring NIV as part of usual clinical care at SCH
* Age 1 month to 16 years.
* Difficulties with current NIV interface
* Only patients that are using NIV for breathing support will be included, ie those with hypoventilation and obstructive sleep apnoea, where the ventilator supports the patient's own breathing.

Exclusion Criteria:

* Families who do not understand written or verbal English where no interpreter is available.
* Children who do not attend with their parent /legal guardian and so are therefore unable to give informed consent.
* Patients deemed too unwell, or unsuitable, by the clinical team
* Patients with adequately functioning NIV interface.
* Patients requiring supplementary medical gases, eg oxygen.
* Patients requiring NIV for rescue breaths will be excluded, ie those with disorders of respiratory control where the ventilator is delivering breaths where the patient has stopped breathing.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient comfort | Until study completion - typically 6 months
  Measured using a investigator devised qualitative diary card
Patient sleep quality | Until study completion - typically 6 months
  Measured using a investigator devised qualitative diary card
Patient skin marking | Until study completion - typically 6 months
  Measured using a investigator devised qualitative diary card
In-patient and home sleep studies | Until study completion - typically 6 months
  Measured using SpO2 and actigraphy monitoring
Mask leak data | Until study completion - typically 6 months
  Measured using ventilator SD card data

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's Hospital, Sheffield, UK, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No